CLINICAL TRIAL: NCT01588691
Title: A Feasibility Study to Examine the Efficacy of C2-C3 Dermatomal Peripheral Nerve Stimulation in Cognitive Improvements Following Persistent Impairment After Traumatic Brain Injury
Brief Title: Traumatic Brain Injury Peripheral Nerve Study
Acronym: TBI
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: CRD-517
Record Dates: First submitted 2012-02-15; First posted 2012-05-01 (Estimated); Last update posted 2019-02-04 (Actual); Status verified 2019-02

CONDITIONS: Traumatic Brain Injury
Keywords: Traumatic Brain Injury
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Low frequency (Active Comparator): Programming parameters with the Eon Mini will be set at a low frequency. Subjects will remain in this group for 3 weeks. If subject cannot tolerate this frequency, he/she will meet with the clinical designee for reprogramming.
  Interventions: Device: Eon-mini IPG (implantable pulse generator)
- High frequency (Active Comparator): Programming parameters with the Eon Mini will be set at a low frequency. Subjects will remain in this group for 3 weeks. If subject cannot tolerate this frequency, he/she will meet with the clinical designee for reprogramming.
  Interventions: Device: Eon-mini IPG (implantable pulse generator)
- No stimulation (Placebo Comparator): Programming parameters will be set to the lowest possible level and minimal power will be generated. Subjects will remain in this group for 3 weeks. If subject cannot tolerate this frequency, he/she will meet with the clinical designee for reprogramming.
  Interventions: Device: Eon-mini IPG (implantable pulse generator)

INTERVENTIONS:
Device: Eon-mini IPG (implantable pulse generator) — programming parameters set at low frequency. Patients will receive this therapy dose for 3 weeks.
  Arms: Low frequency
Device: Eon-mini IPG (implantable pulse generator) — programming parameters set at high frequency. Patients will receive this therapy dose for 3 weeks.
  Arms: High frequency
Device: Eon-mini IPG (implantable pulse generator) — programming parameters set at lowest settings to deliver minimal power. Patients will receive this therapy dose for 3 weeks.
  Arms: No stimulation

SUMMARY:
Peripheral nerve stimulation for the treatment of sequelae due to traumatic brain injury. This study will specifically examine patients with mild traumatic brain injury (TBI) who have persistent cognitive impairments lasting one year or longer. Neuropsychological testing will occur to confirm the diagnosis.

DETAILED DESCRIPTION:
The subject will complete participation in three groups evaluating different programming parameters. After surgery, each subject will be randomized to Group A or Group B. Group C will be completed in the middle followed by the alternate A/B Group. Crossover will occur at 3 week intervals until subjects complete all three groups. During this period, all subjects will receive a subject programmer that will only enable them to activate the "on and off" positions and adjust amplitude within the prescribed range.

After subjects have completed the three pre-defined groups they will select the most effective and comfortable setting continuation of the study. The pulse width and frequency parameters will be set to the optimal settings identified by the subject. Amplitude will be set at a level that produces comfortable paresthesia for the subject.

Subjects will return to the clinic for programming changes post system internalization at 3 weeks, 6 weeks, and 9 weeks. Subjects will receive a PET scan at the 3 and 9 week visit. Additional follow-up evaluations will occur at 12 weeks, 18 weeks, and 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects able to provide informed consent to participate in the study;
2. Subjects between the ages of 18 and 65;
3. Subjects with clear evidence and/or documentation of mild traumatic brain injury as defined by the American Congress on Rehabilitation Medicine (1993):

   * Closed head injury/trauma
   * Score of 13-15 on the Glasgow Coma Scale
   * Documented/witnessed loss of consciousness < 30 minutes post injury
   * Post traumatic amnesia less than 24 hours post injury.
4. Subjects 12 month post-injury with DSM IV diagnosis of Postconcussive Disorder Research Criteria (see Appendix A for detailed definition):

   * Evidence from neuropsychological testing of difficulty in attention or memory
   * Complaints, at baseline, of three or more postconcussive symptoms that have been present at least 3 months.
5. Subject medication that is TBI-related has remained stable for at least 4 weeks prior to baseline data collection;
6. Current medical options have been tried and documented without sufficient improvement in symptom control;
7. Subject agrees not to add or increase any medication throughout the randomization period of the study;
8. Subject is willing to cooperate with the study requirements.

Exclusion Criteria:

1. Subject diagnosed with a terminal disease (ie. cancer, leukemia, or advanced stages of disease resulting in less than 12 months life expectancy);
2. Subject currently participating in another clinical study;
3. Subject with demand-type cardiac pacemakers, an infusion pump or any implantable device (ie. deep brain stimulators, spinal cord stimulators, CSF shunts, aneurism clip and cochlear implants) which may interfere with therapy;
4. Subject with significant depression and/or other significant psychiatric/behavioral problems likely to interfere with study completion or result in addition distress to the subject as determined by a qualified Psychiatrist or psychologist;
5. Subject with an existing medical condition that is likely to require repetitive MRI evaluation in the future (ie. epilepsy, stroke, acoustic neuroma, tumor);
6. Subject with a history of open head trauma;
7. Subject with visual, hearing or motor deficits that impair ability to complete neurocognitive testing;
8. Subject with a history of moderate to severe TBI;
9. Subject with post traumatic seizure disorder;
10. Subject with history of learning disability and/or ADHD
11. Subject with history of chronic headache syndrome prior to post-concussive disorder;
12. Subject is not willing to maintain current TBI-related medication regimen;
13. Female candidates of child bearing potential who are pregnant (confirmed by positive urine/blood pregnancy test), not using adequate contraception (ie. oral contraceptives, injectibles, implants, patches, condoms, barrier methods, spermicides, intrauterine devices, and sterilization), or nursing (lactating) a child.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2011-12; Primary Completion 2014-04 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Reduction in persistent cognitive impairments | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Roni Diaz, Study Director — Abbott Medical Devices
Locations (1):
- Kevin Yoo, MD/Palomar Neurosurgery Ctr, Poway, California, United States